CLINICAL TRIAL: NCT00523146
Title: Treatment of Primary Dysmenorrhea With Kanion Capsule (GF) A Randomized, Double-blind, Placebo-controlled, Repeated-Dose and Multi-Center Clinical Phase II Trial
Brief Title: Treatment of Primary Menstrual Pain With Kanion Capsule
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lianyungang Kanion Group, Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GF-2006-001
Record Dates: First submitted 2007-08-29; First posted 2007-08-31 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2010-02

CONDITIONS: Primary Dysmenorrhea
Keywords: primary dysmenorrhea; Herbal remedy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Kanion Capsule

SUMMARY:
The objectives of this clinical trial are:

* To further study the safety of Kanion Capsule (GF) in primary dysmenorrhea subjects;
* To further evaluate the efficacy of GF in treatment of primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* primary dysmenorrhea

Exclusion Criteria:

* secondary dysmenorrhea

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2007-04; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
pain reduction | 6 months

SECONDARY OUTCOMES:
accompanying symptoms improvement | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jun Shao, Ph.D., Study Chair — Biokey Inc.
Locations (1):
- Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia, United States